CLINICAL TRIAL: NCT05529251
Title: Prospective Therapeutic De-escalation and miRNA-M371 Biomarker Evaluation Phase II Study for Stage IIa/IIb < 3 cm Seminomas
Brief Title: De-escalation Study for Stage IIa/IIb < 3 cm Seminoma
Acronym: EDEN
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Centre Leon Berard (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EDEN (ET21-344)
Record Dates: First submitted 2022-08-26; First posted 2022-09-07 (Actual); Last update posted 2024-01-25 (Actual); Status verified 2024-01

CONDITIONS: Seminoma; Stage II
Keywords: De-escalation; Chemotherapy; Radiotherapy; Carboplatin; Etoposide; Cisplatine; Micro-RNA-M371; PET scan; Overall survival; Biomarker; Efficacy; Progression free rate; Safety; Quality of life
MeSH Terms: conditions — Seminoma

STUDY DESIGN:
Intervention Model Description: * In case of negative week-3 (after 1 EP cyle) PET-scan: Randomization according to 2 arms
    1. Boost of radiotherapy 20 to 30 Gray (Gy) (ARM A)
    2. Carboplatin AUC7 chemotherapy (ARM B)
  * In case of positive week-3 PET-scan: 3 courses of EP chemotherapy (ARM C)
  Parallel observational cohort for patients scheduled to receive standard lumbo-aortic radiotherapy after orchiectomy
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- ARM A (Experimental): RADIOTHERAPY boost 20 to 30 Gy on lymph nodes
  Interventions: Radiation: Radiotherapy boost
- ARM B (Experimental): One cycle of CARBOPLATIN AUC7
  Interventions: Drug: Carboplatin AUC7
- ARM C (Other): 3 cycles of ETOPOSIDE and CISPLATIN
  Interventions: Drug: 3 cycles of EP
- OBSERVATIONAL COHORT (No Intervention): STANDARD RADIOTHERAPY on lymph nodes

INTERVENTIONS:
Radiation: Radiotherapy boost — Radiotherapy boost 20 to 30 Gy, in daily 2 Gy fractions and 5 fractions per week :
  * 20 Gy if no more disease is visible (node < 1 cm in large diameter)
  * 24 Gy for nodes <= 2 cm
  * 30 Gy for nodes > 2 cm
  Arms: ARM A
Drug: Carboplatin AUC7 — Carboplatin at dose (mg) = AUC7 (mg/ml x min) x (DFG ml/min + 25)
  Arms: ARM B
Drug: 3 cycles of EP — 3 Cycles of EP chemotherapy, administred every 3 weeks following standard practice
  Arms: ARM C

SUMMARY:
Phase II, multicenter, prospective, randomized, non-comparative, de-escalation study.

Patients with stage IIa/IIb < 3 cm seminoma histologically proved after orchiectomy will be included in the study and will receive 1 cycle of Etoposide Cisplatine (EP) chemotherapy.

Patients with negative week-3 PET-scan after the EP cycle, will be randomized (1:1 ratio, stratification according to the disease stage (stage IIa versus IIb seminoma)) to receive either radiotherapy (RT) boost on lymph nodes or 1 cycle of carboplatin AUC7 chemotherapy.

Patients with positive week-3 PET-scan will received 3 additional cycles of EP chemotherapy.

In parallel, eligible patients scheduled to receive standard lombo-aortic RT will be registered in an observational cohort.

DETAILED DESCRIPTION:
Stage II seminoma is defined by the presence of retroperitoneal lymph node metastases. It concerns approximately 15% of patients with seminoma. The standard treatment for patients with stage IIa/b seminoma, after orchiectomy, is extended lumbo-aortic/ipsilateral iliac radiotherapy (RT). Performing chemotherapy (CT) with 3 courses of Bleomycin-Etoposide-Cisplatin (BEP) or 4 courses of Etoposide-Cisplatin (EP) is an alternative.

The optimal treatment choice remains controversial. Both treatment modalities are associated with excellent efficacy but also acute and late toxicities. European Society of Medical Oncology (ESMO) guidelines recommended in equal measure CT and RT for stage IIa. A recent systematic review concluded that RT and cisplatin-based combination CT are equally effective in clinical stage IIa/IIb seminoma, with a trend in favor of chemotherapy in stage IIb because of lower relapse rate. However, due to the rarity of stage II seminoma, a sufficiently powered randomized trial comparing radiotherapy with chemotherapy is unlikely to be completed.

De-escalation strategies are required to minimize acute and long-term toxicities while maintaining efficacy. De-escalated treatment for seminoma patients with stage IIb/IIC/III and good prognosis according to International Germ Cell Cancer Collaborative Group (IGCCCG), based on negative PET after 2 cycles of EP chemotherapy, is feasible and safe according to SEMITEP results (cohort 2). In case of negative PET, 1 additional cycle of CT with carboplatin AUC7 was administered.

Furthermore, serum levels of microRNA (miR)-371a-3p (miRNA-M371) have been significantly associated with clinical stage, primary tumor size and response to treatment in testicular germ cell tumors, with sensitivity and specificity higher than those of classic markers (hCGt, LDH). However, further evaluations are needed before modifying clinical practices.

We propose to conduct a multicenter, prospective, randomized, non-comparative, de-escalation phase II study in patients with stage IIa/IIb seminoma < 3 cm, evaluating:

* a more de-escalated CT treatment: 1 cycle of EP followed, in case of negative PET, by either a boost of RT on lymph node or 1 cycle of carboplatin AUC7
* the biomarker miRNA-M371 in therapeutic decision and correlation with PET.

In parallel, eligible patients scheduled to receive standard lombo-aortic RT will be registered in an observational cohort.

ELIGIBILITY:
Inclusion criteria :

1. Age ≥ 18 years on the day of signing informed consent.
2. Primary testicular seminomatous germ cell tumor.
3. Stage IIa/IIb < 3 cm in largest diameter seminoma, histologically proved after orchiectomy.
4. Confirmation of a progressive disease (positive PET scan or increase of lymph nodes size by two successive CT scan).
5. Good prognosis according to IGCCCG and LDH < 2.5 x Upper Limit of Normal (ULN).
6. Normal alpha-fetoprotein (AFP) before and after orchiectomy.
7. No prior treatment with radiotherapy or chemotherapy.
8. Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) ≤ 2.
9. Adequate bone-marrow, hepatic, and renal functions with:

   * Neutrophils ≥ 1.5 x Giga/l, platelets ≥ 100 x Giga/l,
   * Aspartate aminotransferase (AST) and Alanine aminotransferase (ALT) ≤ 1,5 x ULN,
   * Serum creatinine < 140 µmol/l OR calculated clearance > 60 ml/min (using either Cockcroft-Gault formula or Modification of Diet in Renal Disease (MDRD) for > 65 years old),
   * Direct and total bilirubin ≤ ULN.
10. Willingness and ability to comply with scheduled visits, treatment plans, laboratory tests, and other study procedures.
11. Accepting to use effective contraceptive measures or abstain from heterosexual activity, for the course of the study and through 12 months after the last dose of chemotherapy or being surgically sterile. All patients should seek advice regarding cryoconservation of sperm prior treatment initiation because of the possibility of infertility
12. Affiliation to a health insurance.
13. Signed and dated informed consent.

Non-exclusion criteria :

1. Extra-retroperitoneal metastasis on Computed tomography scan (CT scan).
2. Infection by Human Immunodeficiency Virus (HIV), or active infection with the Hepatitis B or C virus.
3. History, within 2 years, of cancer other than seminoma, except for treated skin cancer (basal cell).
4. Uncontrolled or severe cardiovascular pathology.
5. Uncontrolled or severe hepatic pathology.
6. Patient deprived of liberty or requiring tutorship or curatorship.
7. Psychological, physical, sociological, or geographical conditions that would limit compliance with study protocol requirements (at the investigator's discretion).
8. Participation to another clinical trial, except for supportive care trials.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2022-09-06 (Actual); Primary Completion 2025-09-06 (Estimated); Study Completion 2030-09-06 (Estimated)

PRIMARY OUTCOMES:
PFR-36M | Up to 36 months after inclusion
  Progression-free rate at 36 months
  The PFR-36M is assumed to be a random variable following a binomial distribution Bin (n, p) where n is the sample size and p is the true underlying PFR-36M. Conclusions and inferences will be conducted on p. The prior distribution of p (representing the knowledge of the progression-free rate probability prior to observing the data) will be pre-specified. In the absence of a strong idea about the PFR-36M to be observed, a non-informative prior distribution Beta (1,1) will be considered.
  Pr[PFR-36M ≥ 80%] will be expressed in each arm, associated with its 95% credibility interval. A treatment arm will be considered a positive sign for efficacy of de-escalation if there is a high probability that PFR-36M will be higher or equal to 80%: Pr[PFR-36M ≥ 80%] ≥ 90%. It means that if most of the distribution (90% of it) falls to the right hand side of 80%, it indicates that it is very likely that the effect is at least 80%

SECONDARY OUTCOMES:
miRNA-M371 | Up to 5 years
  Serum level of miRNA-M371 as a potential biomarker of response. Association between serum level of miRNA M371 and response to treatments (according to RECIST v1.1) will be evaluated using a non-parametric Wilcoxon Mann and Whitney test and describe with boxplots.
Association of PET scan results and miRNA-M371 rate | Up to 5 years
  Correlation between serum level of miRNA M371 and FDG-PET results (metabolic response) will be evaluated using the Kendall rank correlation and describe graphically.
Overall survival (OS) | Up to 3 years
  The Overall Survival will be defined as the time from date of inclusion to the date of death, from any cause. Patient whose death is not known at the time of analysis will be censored based on the last recorded date on which the patient was known to be alive.
  The Kaplan-Meier (KM) approach will be used to estimate median OS. Median OS as well as Survival rates at specific timepoints will be presented together with their 95% confidence interval (CI).
Quality of life (QoL) | Up to 20 months
  The QoL will be assessed using the EORTC QLQ-C30 questionnaire.
Tolerance to treatment | Up 5 years
  The tolerance to each treatment will be described mainly on the frequency of adverse events (AEs) and their intensity and severity determined using the National Cancer Institute - Common Terminology Criteria for Adverse Events (NCI-CTCAE) grading scale version 5. Descriptive statistics will be provided for characterizing and assessing patient tolerance to treatment.
  AEs will be described and coded, in total and per System Organ Class and Preferred Term with Medical Dictionary for Regulatory Activities (MedDRA) coding

CONTACTS AND LOCATIONS:
Overall Officials: Aude FLECHON, Dr, Principal Investigator — Centre Leon Berard (Lyon, France)
Locations (15):
- France (15):
  - CHU Besançon, Besançon
  - CHU Bordeaux, Bordeaux
  - Centre François Baclesse, Caen
  - Centre Jean Perrin, Clermont-Ferrand
  - Centre Oscar Lambret, Lille
  - CHU de Limoges, Limoges
  - Centre Leon Bérard, Lyon
  - Institut Paoli Calmettes, Marseille
  - Centre Antoine Lacassagne, Nice
  - Hôpital Saint Louis, Paris
  - ICO René Gauducheau, Saint-Herblain
  - Hôpital Foch, Suresnes
  - Institut Universitaire de Cancer de Toulouse (IUCT-O), Toulouse
  - Institut de Cancérologie de Lorraine, Vandœuvre-lès-Nancy
  - Institut Gustave Roussy, Villejuif